CLINICAL TRIAL: NCT00546325
Title: REASURE: The Effect of Rimonabant on HbA1c in Overweight or Obese Patients With Type 2 Diabetes Not Adequately Controlled on 2 Oral Antidiabetic Agents
Brief Title: REASSURE: The Effect of Rimonabant on HbA1c in Overweight or Obese Patients With Type 2 Diabetes Not Adequately Controlled on 2 Oral Antidiabetic Agents
Acronym: REASSURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIMON_L_01661
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Rimonabant
  Interventions: Drug: Rimonabant
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimonabant — White opaque film-coated, for oral administration containing 20 mg of active rimonabant. Once daily before breakfast
  Arms: 1
Drug: Placebo — Matching placebo tablets. Once daily before breakfast
  Arms: 2

SUMMARY:
Primary:

To assess the effects of rimonabant on HbA1c in patients with Type 2 diabetes who are overweight or obese (Body Mass Index (BMI) > 27 kg/m² and BMI < 40 kg/m²), have uncontrolled HbA1c (7.0% - 9.0% inclusive) and are currently on maximal tolerated doses of two Oral Anti Diabetic medications - Metformin (Met) and Sulfonylurea (SU).

Secondary:

To assess the effects of rimonabant on Anthropometric measures, Glucose measures, Lipid measures, Other measures and changes in quality of life

ELIGIBILITY:
List of Inclusion and Exclusion criteria:

Inclusion Criteria:

* History of Type 2 diabetes
* HbA1c between 7% to 9% (inclusive)
* BMI ≥ 27kg/m² and BMI ≤ 40kg/m²
* Currently taking Metformin and Sulfonylurea.

Exclusion Criteria:

* Uncontrolled serious psychiatric illness such as major depression
* Current use of antidepressants
* Severe renal impairment (creatinine clearance less than 30ml/min)
* Severe hepatic impairment known by investigator or Aspartate Aminotransferase and/or Alanine Aminotransferase > 3 times Upper Limit Normal
* Patient treated for epilepsy
* Pregnant or breast-feeding women
* Women of childbearing potential not protected by effective contraception
* Hypersentivity/intolerance to rimonabant or any of the excipents
* Presence of any condition, current or anticipated that in the investigator's opinion would compromise the patient's safety
* Use of insulin for longer than 1 week within 4 weeks prior to screening
* Chronic use of systemic corticosteriods
* Use of glitazone therapy, glucagon-like peptide or dipeptidyl peptidase IV
* History of drug or alcohol abuse wihtin the last three years
* Heart failure class III-IV (New York Heart Association classification)
* Severe hypertension
* Adminstration of the following medications: phentermine, amphetamines, orlistat, sibutramine, herbal remedies
* Use of non-lipid agents known to affect lipid metabolism: retinoids, antiretrovirals, hormone replacement therapy containing estrogens, cyclosporin, thiazolidinediones (glitazones), fish oils, plant sterols
* Use of ketoconazole, itraconazole, ritonavir, clarithromycin, rifampicin, phenytoin, phenobarbitone, carbamazepine or St John's Wort
* Participation in a clinical study within the 4 weeks prior to randomisation
* Patients involved in an existing weight loss program
* Presence of chronic hepatitis
* Use, or misuse, of substances of abuse
* Marijuana or hashish users
* History of gastrointestinal surgery for weight loss purposes or who are scheduled for such surgery within the duration of their expected participation in this study
* History or presence of bulimia or laxative abuse
* Non-English speaking

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Absolute change in HbA1c between both placebo and rimonabant group. | From baseline to week 48
Percentage of participants reaching the treat-to-target objective of HbA1c ≤ 6.5% and ≤ 7.0% | From the beginning to the end of the study
Percentage of participants responding to treatment | From the beginning to the end of study
Rate of asymptomatic, symptomatic, and severe hypoglycaemia | From the beginning to the end of the study
Change in physical examinations, vital signs, laboratory parameters, adverse events | From the beginning to the end of the study

SECONDARY OUTCOMES:
Change in insulin sensitivity, fasting plasma glucose, hypoglycaemia rate. | From the beginning to the end of the study
Change in BMI, waist and hip circumference, waist/hip ratio, weight | From the beginning to the end of the study
Changes in Quality of Life | From the beginning to the end of the study
Change in lipid measures: HDL (High Density Lipoprotein), LDL (Low-Density Lipoprotein), TG (Triglycerides), TC (Total Cholesterol), ApoB (Apolipoprotein B) | From administration of drug till end of study
Change in adiponectin, fasting insulin, Blood Pressure, concomitant medications, health resource use, CRP (C Reactive Protein), ALT (Alanine Aminotransferase), albumin/creatinine ratio | From administration of drug to end of study

CONTACTS AND LOCATIONS:
Overall Officials: David WHEATLEY, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, North Ryde, Australia